CLINICAL TRIAL: NCT06992167
Title: Caregiver Depression in a Low-Resource Setting: Socio-Demographic Predictors of Major Depressive Disorder Among Family Caregivers of Breast Cancer Patients in Pakistan
Status: Completed | Type: Observational
Sponsor: Rahmah Health Foundation (Other)
Responsible Party: Principal Investigator, Muhammad Usman Hashmi, Director, Rahmah Health Foundation
Other Study IDs: RHF-04-2024
Record Dates: First submitted 2025-05-17; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study aims to assess the prevalence of depression among primary caregivers of breast cancer patients within low-resource country like Pakistan. Caregiving for individuals with breast cancer can be physically and emotionally demanding, often leading to psychological distress, including depression. However, there is limited data from low- and middle-income countries, including Pakistan, where caregivers may face additional socioeconomic and systemic burdens. This study seeks to quantify the burden of depression in this population and explore associated sociodemographic and caregiving-related factors. Findings will help inform psychosocial support strategies and interventions to improve caregiver well-being in resource-constrained environments.

ELIGIBILITY:
Inclusion Criteria:

1. Primary caregiver of a patient diagnosed with breast cancer at any stage
2. Male or female caregiver
3. Aged 15 years or older
4. Providing physical, emotional, or financial support to the patient
5. Willing to give informed consent

Exclusion Criteria:

1. Paid caregivers (professional or hired help)
2. Age under 15 years
3. Unwilling to provide consent or participate in the study
4. Incomplete or missing essential data required for analysis

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of primary caregivers of breast cancer patients receiving treatment in public or private healthcare facilities in low-resource settings of Pakistan. Caregivers include family members or individuals who are directly involved in providing physical, emotional, or financial support to the patient.
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of depression among caregivers of breast cancer patients | At a single time point during caregiver recruitment (cross-sectional assessment within 6 months of study initiation)
  Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated screening tool. The PHQ-9 consists of 9 items, each scored from 0 (not at all) to 3 (nearly every day), for a total score range of 0 to 27. Higher scores indicate worse depressive symptoms. Depression severity will be categorized as follows:
  0-4: Minimal
  5-9: Mild
  10-14: Moderate
  15-19: Moderately Severe
  20-27: Severe
  The proportion of caregivers falling into each category will be reported.

CONTACTS AND LOCATIONS:
Locations (4):
- Pakistan (4):
  - Ayub Teaching Hospital, Abbottabad, Pubjab
  - Nishtar Medical University and Hospital, Multan, Punjab Province
  - Jinnah Postgraduate Medical Center, Karachi, Sindh
  - Benazir Bhutto Hospital, Rawalpindi